CLINICAL TRIAL: NCT04013217
Title: A Phase I Study With Expansion Cohorts to Assess the Safety, Tolerability, and Activity of Eribulin ORA in Subjects With Solid Tumors
Brief Title: Evaluate Eribulin ORA in Subjects With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Health Hope Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATX-ERB-001
Record Dates: First submitted 2019-01-09; First posted 2019-07-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eribulin ORA (Experimental): To determine the MTD of Eribulin ORA (oral eribulin mesylate and HM30181A) when administered on Day 1 and Day 8 of a 3 weeks cycle.
  Interventions: Combination Product: Eribulin ORA

INTERVENTIONS:
Combination Product: Eribulin ORA — Oral eribulin mesylate will be supplied as an aqueous solution and HM30181A-UK

SUMMARY:
This is a nonrandomized, open-label, dosed escalation, safety activity, and PK study to determine the MTD and optimal dosing regimen of Eribulin ORA.

DETAILED DESCRIPTION:
This is a multicenter, open-label safety, tolerability, pharmacokinetic, and activity study. Eligible subjects will be adults with advanced solid tumors.

Groups of 3 to 6 subjects will receive a single dose of Eribulin ORA on Day 1 and Day 8 of a 21 day cycle and will be followed for toxicity. If non linearity in PK is observed, additional subjects will be added with study drug administered on Day 1 and 8 once every three weeks cycle. Subjects who tolerate the study drug and have stable disease or better response will be eligible to receive ongoing treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and sign an informed consent form (ICF)
2. Male and female adults, ≥18 years of age
3. Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; subjects enrolling in the dose expansion cohort must have breast cancer or liposarcoma.
4. Must have at least one measurable site of disease as defined as per RECIST v1.1 criteria (dose expansion) or evaluable disease (dose escalation only)
5. Eastern Cooperative Oncology Group (ECOG)2 Performance Status ≤1
6. Adequate hematologic status as demonstrated by not requiring transfusion support or granulocyte-colony stimulating factor (G-CSF) to maintain:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count ≥100 x 109/L
   * Hemoglobin ≥9.0 g/dL
7. Adequate liver function as demonstrated by:

   * Total and direct bilirubin within normal range
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 upper limit of normal (ULN)
   * Gamma-glutamyl transferase (GGT) ≤5 x ULN
   * Alkaline phosphatase ≤3 x ULN or ≤5 x ULN if bone or liver metastasis is present
8. Serum creatinine ≤1.5 x ULN, or estimated creatinine clearance ≥50 mL/min according to the Cockcroft-Gault equation
9. Prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) ≤1.5 x ULN OR if a subject is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of coagulants for 7 days prior to receiving study treatment
10. Subjects receiving warfarin who are otherwise eligible and who may be appropriately managed with low molecular weight heparin, in the opinion of the Investigator, may be enrolled in the study provided they are switched to low molecular weight heparin at least 7 days prior to receiving study treatment.
11. Willing and able to comply with scheduled visits, treatment plan and laboratory tests
12. No concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder
13. Men who are sterile (including vasectomy confirmed by post vasectomy semen analysis) OR agree to use a condom with spermicide and to not donate sperm during the study and for at least 90 days following last dose of Eribulin ORA
14. Female subjects must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using highly effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 90 days after their last dose of assigned study treatment.
15. Subjects who are of childbearing potential must have a negative serum pregnancy test at Screening and within 72 hours before the first dose.

Exclusion Criteria:

1. Subjects who have received recent anti-cancer therapy defined by:

   * Chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies (but excluding nitrosurea, mitomycin-C, targeted therapy) ≤28 days prior to starting study drug, or who have not recovered from side effects of such therapy to Grade 1. Subjects receiving luteinizing hormone-releasing hormone (LHRH) agonists may be considered for enrollment after discussion with the Sponsor.
   * Last administration of nitrosurea or mitomycin-C ≤42 days prior to starting study drug, or who have not recovered from the side effects of such therapy to Grade 1
   * Targeted therapy (eg, sunitinib, sorafenib, pazopanib) ≤14 days prior to starting study drug, or who have not recovered from the side effects of such therapy to Grade 1; or
   * Radiotherapy ≤28 days prior to starting study drug, or ≤14 days prior to starting study drug in the case of localized radiotherapy (eg, for analgesic purpose or for lytic lesions at risk of fracture), or who have not recovered from radiotherapy toxicities to Grade 1.
2. Subject who have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drugs (including gastric bypass surgery and total gastrectomy).
3. Subjects who have undergone major surgery (eg, intra-thoracic, intra-abdominal or intrapelvic), open biopsy or significant traumatic injury ≤28 days prior to starting study treatment, or subjects who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤7 days prior to starting study drug, or who have not recovered from side effects of such procedure or injury
4. Subjects with congenital long QT syndrome
5. Uncontrolled concurrent illness, including but not limited to ongoing or active serious infection requiring systemic antimicrobials (within 14 days prior to first dose), uncontrolled arterial hypertension (>160/100 mm/Hg on antihypertensive medications), chronic pulmonary disease requiring oxygen, known bleeding disorders, uncontrolled endocrine diseases, altered mental status or psychiatric illness/social situations that would limit compliance with protocol requirements.
6. Known or suspected diagnosis of human immunodeficiency virus (HIV) or chronic active Hepatitis B or C, or cirrhosis.
7. Symptomatic or uncontrolled brain metastases requiring current treatment (less than 28 days from last cranial radiation or 28 days from last steroids use).
8. Impaired cardiac function or clinically significant cardiac disease including the following:

   * Clinically significant arrhythmias (except chronic well controlled atrial fibrillation)
   * New York Heart Association (NYHA) Class III or IV congestive heart failure
   * Unstable angina pectoris within the last 6 months
   * Myocardial infarction within the last 6 months
9. Subjects with a healing or open wound
10. Lack of recovery of prior AEs to Grade ≤1 severity (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v4.03)3 (except alopecia or lymphopenia) due to medications administered prior to the first dose of the trial drugs.
11. Any other condition or finding (including social situation) that in the opinion of the Investigator may render the patient at excessive risk for treatment complications or may not be able to provide evaluable outcome information.
12. Pregnant or breast-feeding women
13. Known allergy to any of the formulation components of Eribulin ORA
14. Currently taking following prohibited concomitant medication:

    * Strong cytochrome P450 (CYP) 3A4 inducer (eg, rifampin or St. John's Wort) or a strong CYP3A4 inhibitor (eg, ketoconazole) within 14 days prior to treatment administration
    * Medication known to be strong P-gp inhibitors or inducers. Subjects who are taking such medications but who are otherwise eligible may be enrolled if they discontinue the medication 7 days before dosing and remain off that medication during treatment with Eribulin ORA.
    * An oral medication with a narrow therapeutic index known to be a P-gp substrate (eg, digoxin, dabigatran, colchicine) within 1 day prior to start of Eribulin ORA dosing in the study
    * Drugs known to prolong the QT interval, including Class Ia and III antiarrhythmics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Maximum Tolerated Dose | 3 weeks
  Occurrence of Dose-limiting toxicity (DLT) in all patients who received at lest one dose of Eribulin ORA.
Dose Expansion: Occurrence of Grade 3 and 4 treatment-related adverse | 6 weeks
  Evaluate the occurrence of Grade 3 and 4 treatment-related adverse events to assess the safety of Eribulin IV or Eribulin ORA.

SECONDARY OUTCOMES:
Dose Escalation: Safety | Up to 24 months
  Occurrence of adverse events in all patients who signed the informed consent .
Dose Escalation: Bioavailability | Up to 24 months
  Pharmacokinetic analysis of Area Under the Curve (AUC), Time to Maximum Effect (Tmax), and Peak Plasma Concentration (Cmax) will be done to determine bioavailability of Eribulin IV or Eribulin Ora in all patients who received at least one dose of Eribulin ORA.
Dose Escalation: Tumor Response | up to 24 months
  Evaluate objective tumor response rate for confirmed Partial, Stable, Complete Response, or Progression Disease in all patients who receive at lease one dose of Eribulin IV or Eribulin ORA.

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Health Hope Pharma
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States